CLINICAL TRIAL: NCT04463303
Title: The Role of Lung Ultrasound in The Diagnosis of Weaning -Induced Pulmonary Edema
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ali Ahmed, Lecturer of Internal Medicine, Assiut University
Other Study IDs: LULTRASOUND
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Detecting the Number of B-lines in Lung Ultrasound and Its Accuracy in Diagnosis of Weaning Induced Pulmonary Oedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: patient who will develop weaning induced pulmonary adema
  Interventions: Other: lung ultrasound
- group 2: patient who will nor develop weaning induced pulmonary adema
  Interventions: Other: lung ultrasound

INTERVENTIONS:
Other: lung ultrasound — patient with or without weaning induced pulmonary adema

SUMMARY:
The aim of the work is to

1. Assess the incidence of weaning induced pulmonary adema(WIPO).
2. Assess the risk factors of WIPO.
3. Evaluate the role of lung ultrasound in detecting WIPO during spontenous breathing trial(SBT).
4. Detect the threshold of B-line increase (Delta-B-lines) that provided the best diagnostic accuracy of WIPO.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients on mechanical ventilation who will be suitable for spontaneous breathing trial (SBT).

Exclusion Criteria:

* Patients with poor lung ultrasound window, history of cardiomyopathy, significant valvular disease (aortic or mitral insufficiency of grade ≥ 2, mild or severe aortic and mitral stenosis) will be excluded from the study.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include patients on mechanical ventilation who will be suitable for spontaneous breathing trial (SBT).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
the number of B-lines in lung ultrasound and its accuracy in diagnosis of weaning induced pulmonary oedema | 1 year

IPD SHARING:
Plan to Share IPD: No